CLINICAL TRIAL: NCT01167218
Title: "In-vitro Characterization of Platelet Dysfunction in Common Hematological Disorders Using the Verify Now Assay"
Brief Title: Study to Assess Platelet Dysfunction With Verify Now Assay
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 09318
Record Dates: First submitted 2010-07-19; First posted 2010-07-22 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Platelet Aggregation Defects
Keywords: verify now assay for hematological disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- verify now assay: subjects who have Myelodysplastic syndrome, immune thrombocytopenia, and myeloproliferative disorders with platelet disorders

SUMMARY:
The purpose of this study is to conduct a Verify now assay to detect platelet aggregation defects in patients with Myelodysplastic syndrome(MDS), immune thrombocytopenia purpura (ITP) and myeloproliferative disorders (MPD).

DETAILED DESCRIPTION:
Verify Now is a rapid, simple, point-of service assay to measure platelet aggregation. The verify now assay is designed to assess platelet function based on the ability of activated platelets to bind fibrinogen. It is hoped that this study will detect the subtle platelet functional abnormalities in patients with hematological disorders.

ELIGIBILITY:
Inclusion Criteria

- Patients with common blood disorders such as immune thrombocytopenia purpura(ITP) myelodysplastic syndrome MDS)and myeloproliferative disorders (MPV)

Exclusion Criteria

- Patients with normal platelet counts

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with platelet defects
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2009-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
platelet aggregation defects | one year
  to assess platelet aggregation defects

CONTACTS AND LOCATIONS:
Overall Officials: Nina D'abreo, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital Oncology/Hematology Division, Mineola, New York, United States